CLINICAL TRIAL: NCT05234970
Title: iWellness Study: Evaluation of a CBT Chatbot App to Promote Mental Wellness in Students
Brief Title: iWellness Study to Evaluate a Mental Health App for Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard University (Other)
Responsible Party: Principal Investigator, Leslie Tarver, Principal Investigator, Harvard Medical School (HMS and HSDM)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB21-1024
Record Dates: First submitted 2022-01-21; First posted 2022-02-10 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Depression, Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Participants will be randomly assigned to one of two apps and will be blinded to which is the intervention app and which is the control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator: App 1 Study group (Wysa) (Active Comparator): Wysa App
  Wysa provides free, 24/7, emotional support to users through an app-based AI chatbot system. All Wysa chats are anonymous. The AI-based bot responds to the users' emotions and uses CBT, DBT, meditation, breathing, yoga, motivational interviewing, and micro-actions to help the user manage their emotions and encourage mental well-being. In addition, there are over a hundred AI-guided self-care exercises which are backed by science and handpicked by therapists.
  Interventions: Other: Wysa
- Placebo Comparator: App 2 Study Group (Harvard College Mobile) (Placebo Comparator): Harvard College Mobile App
  "Harvard College Mobile" is an informational app developed by the Harvard University, and is designed to help students navigate resources on campus including professional and peer support groups, but does not allow direct messaging through the app. All Harvard students have full access to the contents of this application.
  Interventions: Other: Harvard College App

INTERVENTIONS:
Other: Wysa — Participants in the intervention arm will be able to log into the Wysa app at any time of day. They can chat with the AI-based bot, Wysa, or choose to complete different self-care exercises. These exercises are grouped into tool packs, which include dealing with relationships, overcoming loneliness, managing mood, among many others. Users can engage in simple, therapeutic exercises including mindfulness and cognitive re-structuring for negative thinking.
  Arms: Active Comparator: App 1 Study group (Wysa)
Other: Harvard College App — Participants in the control arm will be given instructions on how to download and utilize the Harvard College App. Students assigned to this app receive instructions on how to utilize the app to navigate resources on campus to support their mental health including professional and peer support groups and how to make an appointment at the Counseling and Mental Health Services. Participants cannot send messages or share any information through the app.
  Arms: Placebo Comparator: App 2 Study Group (Harvard College Mobile)

SUMMARY:
The study aims to evaluate whether use of a mobile mental health app improves outcomes of depression and anxiety for students.

DETAILED DESCRIPTION:
There is a mental health crisis on college campuses with a growing demand for mental health services and increasing wait times. At the same time, there has been a dramatic surge in the development of mobile mental health apps. Thus, there is an opportunity to leverage these tools to improve mental health services. Our recent pilot study demonstrated the acceptability of using a mental health app to augment college mental health services and the feasibility of a fully digital approach to recruit and randomize students. The findings serve as a proof of concept for a full trial.

Specific Aims:

This study aims to evaluate the effectiveness of a mental health app to improve symptoms of depression and anxiety for students compared to treatment as usual.

In our pilot study, the investigators limited recruitment to students waiting for an initial appointment at Harvard University Health Services (HUHS) Counseling and Mental Health Services (CAMHS). In this trial, the investigators will broaden enrollment to include students seeking care at CAMHS as well as students who are not currently enrolled in treatment but who could benefit from additional mental health support.

In addition, in the full trial, the investigators will explore mediators of change, including perceived stress and isolation, through which a Cognitive Behavioral Therapy (CBT)-based Chatbot app ("Wysa") may contribute to improvement in depression and anxiety among students.

This will also involve exploring possible moderators of the effect such as students' demographic characteristics, concurrent or previous mental health treatment, and degree of usage of the mobile app.

The mobile mental health app will not be offered as a replacement for treatment at HUHS CAMHS but as a way of offering initial support and a potential gateway to seeking further treatment. In addition, the app is intended to promote mental wellness as using the app will help give students skills that may prevent them from needing further mental health treatment. For those with active symptoms, it is meant to increase students' interest in engaging with mental health services.

This study will make a significant and novel contribution to research in college mental health regarding the effectiveness of mobile mental health applications in the college population. Additionally, it will help provide understanding of the mediators of this effect and whether an innovative tool such as a CBT chatbot app can be used to promote mental wellness, prevent worsening mental health symptoms and increase uptake with other mental health related services for students who are not engaged in traditional treatment.

The investigators propose to address the following aims:

Aim 1: Evaluate the use of a CBT-based mobile Chatbot app ("Wysa") to improve outcomes of depression and anxiety for students compared to treatment as usual as measured by improvement in PHQ-9 and GAD-7 scores.

Hypothesis 1: Participants randomly assigned to the intervention will be more likely to report improved anxiety and depression outcomes, assessed after the intervention, compared to the participants randomly assigned to the control group (Cohen d = 0.4).

Aim 2: Assess the potential mediators of change for a CBT-based Chatbot app ("Wysa") to improve depression and anxiety.

Hypothesis 2: Perceived stress and social isolation will be identified as potential mediators of the relationship between the intervention and depression and anxiety.

Background and Significance

Untreated or under-treated depression and anxiety in college-age students has tremendous costs for the individual, the larger community and society at large, with the fatal outcome of suicide leading to devastating consequences for college communities. The frequency that students report having seriously considered suicide has increased by almost 40% in the last five years and the demand for counseling services has also grown five times faster than average student enrollment. Technological innovations such as mobile apps hold promise to improve access to care, allow students to seek care in a way that is potentially more comfortable for them, and to alleviate demand on over-burdened service centers. However, there is limited evidence on the effectiveness, feasibility of use and mechanisms by which these mobile platforms may improve mental health outcomes. Consequently, there is a pressing need to further research the use of mobile apps in this population to improve care and inform novel treatment approaches.

Considering the ubiquity of mobile phone usage in this population-98% of young adults aged 18-29 own a smartphone -there is significant interest in the use of mobile phone apps as an alternate care delivery platform. Additionally, the number of mobile mental health apps is exponentially growing with currently thousands of mental health apps available. Mobile apps have the potential to reach people outside of the traditional care model and allow people to use these tools when they need them, and as often as they like without having to wait for a mental health professional. Additionally, mobile health applications offer advantages such as continuous availability and immediate support, anonymity, customizable content and self-guided treatment approaches. These tools have also been seen as ways to increase service capacity and efficiency, reduce other barriers to face-to-face help seeking such as stigma and shame, and may be particularly well suited to young people who may be more accepting of technological approaches.

However, the evidence base for the efficacy of digital technologies for the mental health of college students remains unclear and research is significantly lagging behind app development. A systematic review found that even though many studies found that digital mental health interventions were effective, about half of the studies failed to present any usability or acceptability outcomes. They found that further research on user experience and engagement would be vital to the success of digital mental health interventions on college campuses. Furthermore, another study found that the largest problem for top-ranked apps for depression was attrition; the value of an AI-based chatbot lies in its ability to respond real-time to a user's inputs. Lastly, a scoping systematic review focused specifically on mental digital health platforms for university students found that students worldwide were prepared to engage with digital mental health interventions but placed a high emphasis on a need for reliable devices handling their sensitive data.

This study seeks to advance the initial findings from our pilot study and address current gaps in the literature. By selecting an interactive, AI-chatbot app, our study also aims to explore the role of an innovative approach to providing mental health resources and improving mental wellness for students.

Research Design

This is a randomized controlled trial conducted fully digitally to evaluate the effectiveness of a mobile chatbot app to alleviate symptoms of depression and anxiety in students.

Methods

Recruitment and Screening This trial will include a broad recruitment strategy with a focus on mental health promotion. Students who are both engaged in treatment at HUHS and those who are not engaged in treatment will be allowed to participate.

The recruitment strategy is detailed below:

HUHS/CAMHS:

Students visiting the HUHS website or the CAMHS website will be able to view information about the study and a link which will direct them to the iWellness Study website in order to enroll.

Students who seek care at HUHS CAMHS for symptoms of depression and anxiety will be offered the option to participate in the study when registering for an initial assessment at HUHS CAMHS. Students will be directed to the study website to view information about the study and a link to complete an enrollment eligibility survey.

Other recruitment efforts:

* Harvard graduate students who have completed a mental wellness survey as part of the Graduate Student Mental Health Initiative led by Dr. Paul Barreira would be invited to participate in this study after completing the survey by clicking on the link to enroll. The graduate wellness survey is accessible and distributed to graduate students in departments who agree to participate.
* Students will be able to obtain information about the study through campus outreach efforts for mental health promotion including the college and graduate/professional schools.
* Students will also be able to obtain information through relevant campus organizations and campus resource centers. Students would be directed to study information on the HUHS website.

Sample size: By targeting a broader population for recruitment our goal will be to recruit approximately 250-300 students in the study over approximately a 3-month enrollment period.

This is estimated based on data from our recruitment sources including students making new appointments at HUHS CAMHS, visiting the HUHS website, and Harvard graduate students who complete a mental health screening who would all be invited to participate in the study.

This sample size would allow us to obtain 0.80 power to detect significant improvement (Cohen d = 0.4) and significance 0.05.

Baseline Assessment and Group Assignment

Once a participant is recruited, they will go through the same enrollment process as in the pilot study in which they will be directed to the study enrollment website where interested participants will complete a survey to determine eligibility including information about basic demographics and mobile device ownership. Those meeting basic eligibility requirements will also complete screening using the Patient Health Questionnaire - 9 (PHQ-9) and the Generalized Anxiety Disorder 7-item scale (GAD-7) to determine final eligibility. If eligible, participants will agree to participate via an electronic consent form.

In order to test the possible mediator of change, participants will also be asked to fill out a baseline assessment of perceived stress using the Perceived Stress Scale and isolation using the Hughes Loneliness Scale.

Participants will then be randomly assigned to either the Wysa intervention app or the Harvard College Mobile app and given instructions on how to download their assigned app. Participants from both groups will continue to use their assigned app for 8 weeks after enrollment. Participants will receive a secure Qualtrics survey via email at 2-weeks, 4-weeks and 8-weeks. The endpoint of the study will be 8-weeks after enrollment. At the 8-week endpoint, participants will again receive a secure survey including the PHQ-9, GAD-7, Perceived Stress Scale, and the Hughes Loneliness Scale and questions about their satisfaction with the app and their overall care.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be required to be at 18 years or older
* Own a smartphone with Wi-Fi or 3G/4G capabilities
* Current student at Harvard University
* A PHQ-9 score of 5 or greater (indicating mild symptoms of depression or greater), or a score of 2 or greater on PHQ item 10 (indicating that they felt disabled in their life because of their mood) or a GAD-7 score of 8 or greater (indicating mild symptoms of anxiety or greater) will be required for enrollment.

Exclusion Criteria:

* Those who score less than 5 on PHQ-9 or less than 8 on the GAD-7 during study screening will be excluded from the study.
* Anyone who indicates thoughts of harm to themselves or others (PHQ-9 item 9 score > 0) during initial screening will be excluded from participation in the study.
* Participants with a PHQ-9 Q9 suicide item score > 0 will receive an automated notification that they are not eligible to participate in the study and that they should call the Harvard Counseling and Mental Health Services 24/7 line. Study staff will also inform Chief of HUHS CAMHS to reach out to the participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Depression - Patient Health Questionnaire - 9 (PHQ-9) | 8 weeks
  PHQ-9: A 9-question multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression.
  Scoring: Scoring: 0-3 Scale for each item; 0 Not at all; 3 Nearly every day
  The nine item version of the PHQ-9 was designed to facilitate the recognition and diagnosis of depression in primary care patients. It can be used to monitor change in symptoms over time and provides a depression severity index score as follows:
  0-4 None 5-9 Mild 10 - 14 Moderate 15 - 19 Moderately Severe 20 - 27 Severe The recommended cut-off for the PHQ-9 severity index is a score of 9. Anyone who scores 10 or above can be considered to be suffering from clinically significant symptoms of depression.
Anxiety - Generalized Anxiety Disorder 7-item scale (GAD-7) | 8 weeks
  GAD-7: A diagnostic self-report 7-item scale for screening, diagnosis, and severity assessment of generalized anxiety disorder.
  Scoring: 0-3 Scale for each item; 0 Not at all; 3 Nearly every day
  The index scores are as follows:
  0-4 None 5-10 Mild Anxiety 11 - 15 Moderate Anxiety 15 - 21 Severe Anxiety
  The recommended cut off for the GAD-7 severity index is a score of 7. Anyone who scores 8 or above can be considered to be suffering from clinically significant anxiety symptoms.

SECONDARY OUTCOMES:
Perceived Stress - Perceived Stress Scale (PSS) | 8 weeks
  PSS: A psychological instrument for measuring the perception of stress by asking about feelings and thoughts during the last month.
  PSS scores are obtained by reversing responses (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) to the four positivelystated items (items 4, 5, 7, & 8) and then summing across all scale items. A short 4 item scale can be made fromquestions 2, 4, 5 and 10 of the PSS 10 item scale.
Loneliness - Hughes Loneliness scale | 8 weeks
  Hughes Loneliness scale: This is a scale used to assess feelings of loneliness or social isolation. The Three-Item Loneliness Scale is a questionnaire developed from the Revised UCLA Loneliness Scale.
  Each question is rated on a 3-point scale:
  1. = Hardly Ever
  2. = Some of the Time
  3. = Often.
  Scoring: All items are summed to give a total score. Higher scores indicate greater degrees of loneliness.

CONTACTS AND LOCATIONS:
Overall Officials: Giang Nguyen, MD, Study Director — Harvard University
Locations (1):
- Harvard University Health Services, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aboujaoude E, Salame W, Naim L. Telemental health: A status update. World Psychiatry. 2015 Jun;14(2):223-30. doi: 10.1002/wps.20218. PMID 26043340
- [Background] Andrews G, Cuijpers P, Craske MG, McEvoy P, Titov N. Computer therapy for the anxiety and depressive disorders is effective, acceptable and practical health care: a meta-analysis. PLoS One. 2010 Oct 13;5(10):e13196. doi: 10.1371/journal.pone.0013196. PMID 20967242
- [Background] Anthes E. Mental health: There's an app for that. Nature. 2016 Apr 7;532(7597):20-3. doi: 10.1038/532020a. No abstract available. PMID 27078548
- [Background] Arean PA, Hallgren KA, Jordan JT, Gazzaley A, Atkins DC, Heagerty PJ, Anguera JA. The Use and Effectiveness of Mobile Apps for Depression: Results From a Fully Remote Clinical Trial. J Med Internet Res. 2016 Dec 20;18(12):e330. doi: 10.2196/jmir.6482. PMID 27998876
- [Background] Center for Collegiate Mental Health (CCMH). 2016 Annual Report. Publication No. STA 17-74. January, 2017.
- [Background] Center for Collegiate Mental Health (CCMH). 2020 Annual Report. Publication No. STA 21-045. January, 2021.
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Firth J, Torous J, Nicholas J, Carney R, Pratap A, Rosenbaum S, Sarris J. The efficacy of smartphone-based mental health interventions for depressive symptoms: a meta-analysis of randomized controlled trials. World Psychiatry. 2017 Oct;16(3):287-298. doi: 10.1002/wps.20472. PMID 28941113
- [Background] Grist R, Porter J, Stallard P. Mental Health Mobile Apps for Preadolescents and Adolescents: A Systematic Review. J Med Internet Res. 2017 May 25;19(5):e176. doi: 10.2196/jmir.7332. PMID 28546138
- [Background] Montagni I, Tzourio C, Cousin T, Sagara JA, Bada-Alonzi J, Horgan A. Mental Health-Related Digital Use by University Students: A Systematic Review. Telemed J E Health. 2020 Feb;26(2):131-146. doi: 10.1089/tmj.2018.0316. Epub 2019 Mar 19. PMID 30888256
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Lattie EG, Adkins EC, Winquist N, Stiles-Shields C, Wafford QE, Graham AK. Digital Mental Health Interventions for Depression, Anxiety, and Enhancement of Psychological Well-Being Among College Students: Systematic Review. J Med Internet Res. 2019 Jul 22;21(7):e12869. doi: 10.2196/12869. PMID 31333198
- [Background] Mistler, et al. Association for University and College Counseling Center Directors Annual Survey, 2012.
- [Background] Mohr DC, Burns MN, Schueller SM, Clarke G, Klinkman M. Behavioral intervention technologies: evidence review and recommendations for future research in mental health. Gen Hosp Psychiatry. 2013 Jul-Aug;35(4):332-8. doi: 10.1016/j.genhosppsych.2013.03.008. Epub 2013 May 8. PMID 23664503
- [Background] Pew Research Center. Mobile Fact Sheet. April 7, 2021. < https://www.pewresearch.org/internet/fact-sheet/mobile/>
- [Background] Qu C, Sas C, Dauden Roquet C, Doherty G. Functionality of Top-Rated Mobile Apps for Depression: Systematic Search and Evaluation. JMIR Ment Health. 2020 Jan 24;7(1):e15321. doi: 10.2196/15321. PMID 32012079
- [Background] Rosenberg, Morris. 1989. Society and the Adolescent Self-Image. Revised edition. Middletown, CT: Wesleyan University Press.
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Anderson M. Technology device ownership. Washington, DC: Pew Research Center; 2015.